CLINICAL TRIAL: NCT07251335
Title: Melanoma of the Skin and Exposure to Solar Ultraviolet Radiation at Work in Modena Territory: a Case-control Study to Promote an Active Search and Prevention of Occupational Diseases Based on Recent INAIL Criteria
Acronym: Mesur
Status: Recruiting | Type: Observational
Sponsor: University of Modena and Reggio Emilia (Other)
Responsible Party: Principal Investigator, Alberto Modenese, Director of the Occupational Medicine Residency Program, Department of Biomedical, Metabolic and Neural Sciences University of Modena & Reggio Emilia (UniMoRe), University of Modena and Reggio Emilia
Other Study IDs: FAR_438_2024; GRANT_NUMBER: PRJ-0532 FAR2024 (Other Grant/Funding Number: University of Modena and Reggio Emilia - Finanziati FAR Progetti 2024 - Linea FOMO)
Record Dates: First submitted 2025-11-18; First posted 2025-11-26 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-10

CONDITIONS: Skin Melanoma; Cutaneous Melanoma
Keywords: Skin melanoma; Cutaneous Melanoma; Occupational Exposure; Solar Ultraviolet Radiation; Outdoor Workers; Case-Control Study; Occupational Disease; Skin Cancer; Cumulative Sun Damage; Lentigo Maligna Melanoma; Occupational Health; Dermatology; Italy; Occupational Medicine
MeSH Terms: conditions — Melanoma; Occupational Diseases; Skin Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Participants in this group are patients recruited from the Dermatology Clinic who have received a new, histopathologically confirmed diagnosis of skin melanoma.
- Controls: Participants in this group are patients recruited from the same Dermatology Clinic who have been screened negative for melanoma. These controls are matched to the cases based on similar age and gender.

SUMMARY:
The goal of this observational study is to learn about the link between work-related sun exposure and a specific type of skin cancer called melanoma in people living in the Modena area, Italy.

The main questions it aims to answer are:

* Is there a connection between working outdoors and developing types of melanoma that are linked to long-term sun exposure?
* Can we use recent criteria from the Italian workers' compensation authority (Istituto Nazionale per l'Assicurazione contro gli Infortuni sul Lavoro, INAIL) to better identify and report these melanomas as occupational diseases?

Participants in this study will:

* Be patients of the Modena University Hospital Dermatology Clinic who are already undergoing a skin biopsy for a suspected lesion.
* Take part in a one-time interview with a trained healthcare worker.

Answer questions about their:

* Job history and specific work locations (to calculate local UVR exposure).
* Sun exposure habits at work and in their free/holiday time.
* Use of sun protection (e.g., sunscreen, protective clothing).
* Use of tanning beds.
* Natural skin color and tendency to sunburn (and other elements to determine their specific skin phototype).
* Other personal and family health factors.

Researchers will compare two groups:

* Cases: 120 participants who are diagnosed with melanoma after the biopsy.
* Controls: 180 participants who screened negative for melanoma but may show another skin condition.

By comparing these groups, researchers aim at better understanding the role of outdoor work as a risk factor for specific melanoma subtypes. For participants diagnosed with a melanoma that is likely linked to their job, the study team will promote its reporting as an occupational disease.

DETAILED DESCRIPTION:
This is a monocentric, observational, case-control study conducted at the Dermatology Clinic of the University Hospital of Modena (Azienda Ospedaliero-Universitaria di Modena), Italy.

Background and Rationale:

Skin melanoma is a significant public health concern. While its link to solar ultraviolet radiation (UVR) is established, the specific role of occupational (long-term, cumulative) exposure, as opposed to recreational (intermittent, intense) exposure, is still a subject of detailed investigation. In the period 2008-2014, skin melanoma was included in List 2 (limited probability of occupational origin) of diseases to be mandatorily reported as "occupational" by physicians (Italian law DPR 1124/1965) for the exposure agent "solar radiation". After 2014, it was removed from that list, partly due to evolving scientific evidence suggesting that UV-related malignant melanoma was more strongly related to a pattern of solar ultraviolet radiation exposure typically associated with leisure time activities rather than occupational outdoor activities, especially during childhood and adolescence. Recent classifications by the World Health Organization (WHO) now distinguish melanoma subtypes based on their association with cumulative solar damage (CSD). This is a crucial development, as occupational outdoor activity is a primary factor associated with cumulative sun damage. A joint WHO/International Labour Organization (ILO) meta-analysis found a significantly increased risk for one specific CSD-related subtype, Lentigo Maligna Melanoma, in outdoor workers. In line with this, the Italian National Institute for Insurance against Accidents at Work (Istituto Nazionale per l'Assicurazione contro gli Infortuni sul Lavoro, INAIL) has recently proposed new criteria for recognizing specific CSD-related melanomas as occupational diseases in this worker population.

This study aims to apply these novel criteria in a clinical setting to investigate the association between occupational UVR exposure and CSD-related melanoma subtypes.

Study Objectives:

- The primary objective is to evaluate the association between occupational solar UVR exposure and the risk of developing melanoma, with a specific focus on subtypes related to cumulative solar damage (CSD).

Secondary objectives include:

* Comparing occupational and recreational UVR exposure patterns between melanoma cases and controls.
* Correlating melanoma subtypes (CSD-related vs. non-CSD-related) and their body location with specific UVR exposure histories.
* Applying the recent INAIL criteria to identify cases of melanoma that qualify for reporting as occupational diseases.
* Quantitatively estimating individual occupational UVR exposure levels by applying a validated European job-exposure matrix (JEM) developed by Würtz et al. in 2025.
* Calculating and comparing an individualised melanoma risk score for each participant, based on established non-occupational risk factors, according to the model developed and externally validated by Fortes et al. in 2010.
* Analysing the relationship between quantitative occupational UVR exposure and the individualised melanoma risk score.

Study Population and Recruitment:

The study population will consist of patients referred to the Dermatology Clinic for examination of suspicious skin lesions. All enrolled participants will provide written informed consent.

Cases: Approximately 120 adult patients (≥18 years) with a new, histopathologically confirmed diagnosis of cutaneous melanoma.

Controls: Approximately 180 adult patients (≥18 years) who undergo a dermatological screening for a suspicious lesion, but for whom the result of the screening is negative for melanoma. These controls will be matched to cases based on similar age and gender to minimize confounding.

Methods:

Data Collection: After enrolment, all participants (cases and controls) will undergo a single, structured interview conducted by trained healthcare personnel (e.g., resident physicians). The interview will use a detailed questionnaire designed specifically for this study based on a comprehensive literature review.

Questionnaire Content: The questionnaire will collect data on:

* Socio-demographics and general information: Age, gender, country of birth, smoking habits, physical characteristics linked to determine phototype, ease of sunburn, residential history.
* Dermatological anamnesis: Skin melanoma diagnosis, type of melanoma, location, past diagnosis of skin melanoma(ta) and location, past diagnosis of non-melanoma(ta) skin cancers, family history of melanoma and other skin cancers, presence and number of lentigines in sun-exposed and non-sun-exposed areas, presence and number of nevi on the arms and on the rest of the body; history of prolonged treatments with immunosuppressors; use of tanning beds.
* Occupational History: A detailed, chronological work history. For every job (classified according to the international ISCO-88 classification), the specific job duties, the general company activities, and the country and region (for latitude-based UV index assessment) will be required. If possible, specific dates of job start and job end will be collected, as well as the frequency of use of UVR protective measures (clothing, hat, or sun creams).
* Extra-work solar exposure: The study will investigate the habits of staying outside, frequency of sunburn, going to the sea or to high mountains, and the use of sun protection creams, hats, or UV protective clothing. Data will be separated for holiday time versus free/leisure time, and further divided for the age periods 0-20 and ≥21 years.

Data Management and Analysis:

* Data Handling: All collected data will be anonymized and stored in a secure electronic database (RedCap).
* Exposure Assessment: An expert assessment, guided by a Job Exposure Matrix developed from the EU-funded EPHOR project, will be used to categorize participants' cumulative occupational UVR exposure.
* Statistical Analysis: Standard descriptive statistics will characterize the study population. The association between UVR exposure (both occupational and recreational) and other risk factors for melanoma will be assessed by calculating Odds Ratios (OR) with 95% confidence intervals using multivariate regression analysis. Subgroup analyses will be performed based on melanoma subtype and tumour location. Statistical software such as STATA or SPSS will be used.

Quality Assurance:

The study protocol, including the questionnaire and data management plan, will be standardized. Interviewers will receive specific training to ensure consistent data collection. Data entry will include range and consistency checks to ensure quality.

Ethical Considerations:

The study will be conducted after approval from the relevant Ethical Committee of the University Hospital of Modena. Participation is voluntary, and participants may withdraw at any time without affecting their medical care. For outdoor workers diagnosed with a CSD-related melanoma located on sun-exposed skin, the study procedure includes assistance in reporting the disease to INAIL as a potential occupational illness, as per current Italian recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Be a patient of the Dermatology Clinic at the University Hospital of Modena.
* Be 18 years of age or older.
* Have undergone a dermatological screening for a suspected skin lesion.
* Be able to understand and sign an informed consent form in italian language.

Exclusion Criteria:

* Be under 18 years of age.
* Have cognitive impairment that prevents providing reliable answers to the interview or recalling past exposures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be selected from the patient cohort attending the Dermatology Clinic of the University Hospital of Modena (Azienda Ospedaliero-Universitaria di Modena), Italy. This clinic serves a large number of citizens from the Modena province and surrounding areas each year, providing a representative sample for investigating skin cancer. Participants will be identified from among those referred to the clinic for the examination and diagnosis of suspicious pigmented skin lesions.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-07-07 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Association between occupational solar UVR exposure and melanoma diagnosis. | The Odds Ratio will be calculated and assessed once, at the end of the data collection and analysis phase (at the end of the study).
  The strength of the association will be measured by calculating the Odds Ratio (OR) for melanoma in participants with a history of occupational solar UVR exposure compared to those without, using multivariate analysis.

SECONDARY OUTCOMES:
Association stratified by melanoma subtype. | Through study completion, up to 24 months.
  Analysis of the association (measured by Odds Ratios) between occupational solar UVR exposure and specific melanoma subtypes, classified according to the 2018 WHO criteria (e.g., high Cumulative Solar Damage (CSD) subtypes like Lentigo Maligna Melanoma vs. low-CSD subtypes vs. non-solar subtypes).
Association stratified by tumour location. | Through study completion, up to 24 months.
  Analysis of the association (measured by Odds Ratios) between occupational solar UVR exposure and melanoma occurring on chronically sun-exposed body sites versus less exposed or non-exposed sites.
Proportion of melanoma cases reported as occupational diseases. | Through study completion, up to 24 months.
  The number and proportion of melanoma cases that meet the recent INAIL criteria for being reported as an occupational disease due to solar UVR exposure. This applies to outdoor workers diagnosed with a CSD-related melanoma located on photo-exposed body regions.
Quantitative occupational UVR exposure level computation. | Through study completion, up to 24 months.
  The cumulative occupational solar UVR exposure level for each participant with a history of outdoor work will be estimated using the quantitative European job-exposure matrix (JEM) developed by Würtz et al. Exposure will be expressed in Standard Erythemal Doses (SED).
Individualised melanoma risk score computation. | Through study completion, up to 24 months.
  A quantitative melanoma risk score will be calculated for each participant (both cases and controls) using a risk prediction model developed by Fortes et al. in 2010. This model incorporates known non-occupational risk factors such as skin phototype, hair and eye colour, freckling, family history of melanoma, number of common nevi, and history of sunburns.
Association between quantitative occupational UVR exposure and melanoma risk score. | Through study completion, up to 24 months.
  Analysis of the relationship between the quantitatively estimated occupational UVR exposure (from the JEM) and the individualised melanoma risk score, to investigate potential interactions or confounding.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Modenese, MD. PhD, Principal Investigator — University of Modena and Reggio Emilia; Francesca Farnetani, MD, Study Chair — University of Modena and Reggio Emilia; Paola Ferri, MSc, Study Director — University of Modena and Reggio Emilia; Sergio Rovesti, MD, Study Director — University of Modena and Reggio
Locations (1):
- Dipartimento di Scienze Biomediche, Metaboliche e Neuroscienze, Modena, Mo, Italy

IPD SHARING:
Plan to Share IPD: No
The Individual Participant Data (IPD) collected for this study contains detailed and sensitive personal information, including medical histories, occupational records, and lifestyle factors. To ensure the confidentiality and privacy of our participants in compliance with stringent EU and Italian data protection regulations (GDPR), the data will not be made publicly available. The data will be kept securely within the institutional responsibility of the University of Modena and Reggio Emilia for the purposes outlined in this protocol.

REFERENCES:
- [Result] DECRETO DEL PRESIDENTE DELLA REPUBBLICA 30 giugno 1965, n. 1124. Testo unico delle disposizioni per l'assicurazione obbligatoria contro gli infortuni sul lavoro e le malattie professionali. GU n.257 del 13-10-1965 - Suppl. Ordinario (Ultimo aggiornamento all'atto pubblicato il 18/11/2023)
- [Result] Armstrong BK, Cust AE. Sun exposure and skin cancer, and the puzzle of cutaneous melanoma: A perspective on Fears et al. Mathematical models of age and ultraviolet effects on the incidence of skin cancer among whites in the United States. American Journal of Epidemiology 1977; 105: 420-427. Cancer Epidemiol. 2017 Jun;48:147-156. doi: 10.1016/j.canep.2017.04.004. Epub 2017 May 3. PMID 28478931
- [Result] Elder DE, Bastian BC, Cree IA, Massi D, Scolyer RA. The 2018 World Health Organization Classification of Cutaneous, Mucosal, and Uveal Melanoma: Detailed Analysis of 9 Distinct Subtypes Defined by Their Evolutionary Pathway. Arch Pathol Lab Med. 2020 Apr;144(4):500-522. doi: 10.5858/arpa.2019-0561-RA. Epub 2020 Feb 14. PMID 32057276
- [Result] Inail - Sovrintendenza sanitaria centrale: Patrizio Rossi, Grazia Genga Mina. Il melanoma cutaneo professionale da radiazioni solari aspetti d'interesse medico-legale e prevenzionali. ISBN 978-88-7484-825-6
- [Result] Chiossi R. Melanoma, 270 diagnosi in un anno. Il 70% scoperto in fase precoce. Gazzetta di Modena, 23/5/2023, available online: https://www.gazzettadimodena.it/modena/cronaca/2023/05/23/news/melanoma-270-diagnosi-in-un-anno-il-70-scoperto-in-fase-precoce-1.100310134
- [Result] Paulo MS, Adam B, Akagwu C, Akparibo I, Al-Rifai RH, Bazrafshan S, Gobba F, Green AC, Ivanov I, Kezic S, Leppink N, Loney T, Modenese A, Pega F, Peters CE, Pruss-Ustun AM, Tenkate T, Ujita Y, Wittlich M, John SM. WHO/ILO work-related burden of disease and injury: Protocol for systematic reviews of occupational exposure to solar ultraviolet radiation and of the effect of occupational exposure to solar ultraviolet radiation on melanoma and non-melanoma skin cancer. Environ Int. 2019 May;126:804-815. doi: 10.1016/j.envint.2018.09.039. Epub 2019 Feb 18. PMID 30792021
- [Result] Gobba F, Dall'Olio E, Modenese A, De Maria M, Campi L, Cavallini GM. Work-Related Eye Injuries: A Relevant Health Problem. Main Epidemiological Data from a Highly-Industrialized Area of Northern Italy. Int J Environ Res Public Health. 2017 Jun 6;14(6):604. doi: 10.3390/ijerph14060604. PMID 28587288
- [Result] Modenese A, Loney T, Ruggieri FP, Tornese L, Gobba F. Sun protection habits and behaviors of a group of outdoor workers and students from the agricultural and construction sectors in north-Italy. Med Lav. 2020 Apr 30;111(2):116-125. doi: 10.23749/mdl.v111i2.8929. PMID 32352425
- [Result] Modenese A, Farnetani F, Andreoli A, Pellacani G, Gobba F. Questionnaire-based evaluation of occupational and non-occupational solar radiation exposure in a sample of Italian patients treated for actinic keratosis and other non-melanoma skin cancers. J Eur Acad Dermatol Venereol. 2016 Apr;30 Suppl 3:21-6. doi: 10.1111/jdv.13606. PMID 26995019
- [Result] Wurtz ET, Pugdahl K, Fenger-Gron M, Berglind IA, Cherrie MPC, Dahlman-Hoglund A, Grandahl K, Macan J, Modenese A, Noto H, Solovieva S, Straif K, Wittlich M, Connemann S, Heepenstrick T, Philipsen PA, Westerhausen S, Ge CB, Hansen J, Peters CE, Mehlum IS, Schlunssen V, Kolstad HA. A quantitative solar ultraviolet radiation job-exposure matrix for Europe. Ann Work Expo Health. 2025 Apr 24;69(4):415-428. doi: 10.1093/annweh/wxaf011. PMID 40056460